CLINICAL TRIAL: NCT05803759
Title: The Effects of Dietary Supplementation Allicor on the Effectiveness of Treatment of Patients After Coronary Arteria Revascularization
Brief Title: The Effects of Allicor on Patients After Coronary Arteria Revascularization Treatment
Acronym: TEA-CART
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAR-AL-CAR
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Ischemia; Coronary Artery Bypass Grafting; Coronary Arteriosclerosis; Percutaneous Coronary Revascularization
Keywords: Inflammation; Allicin; Mitochondrial Genome
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allicor (Active Comparator): Dietary Supplement: Allicor 150 mg capsule by mouth two times a day
  Interventions: Dietary Supplement: Allicor
- Placebo (Placebo Comparator): Placebo capsule manufactured to mimic Allicor 150 mg capsule by by mouth two times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Allicor — Each capsule contains 150 mg dried garlic powder
  Other Names: 150 mg capsules of dried dried garlic powder
  Arms: Allicor
Drug: Placebo — Capsules manufactured to mimic Allicor 150 mg capsules
  Other Names: Allicor immitation
  Arms: Placebo

SUMMARY:
Coronary revascularization interventions such as coronary artery bypass graft (CABG) and percutaneous coronary intervention (PCI) are the standard of surgical treatment of patients with myocardial ischemia. However, up to 30% of patients experience complications of varying degrees within 12 months after the revascularization, or need for second intervention. Thus, it is necessary to search for additional approaches to the postoperative treatment of patients in order to improve the long-term results of revascularization treatment. Substances of natural origin with an anti-atherosclerotic effect have a good potential. These substances, as dietary supplements, can be taken by patients for a long time in conjunction with other prescribed medicines and treatments. Another valuable direction of investigations is the search for predictors of long-term cardiovascular complications after revascularization, which can be markers of inflammation and heteroplasmy levels of the patient's mitochondrial genome.

The purpose of this study is to determine whether the intake of dietary supplement Allicor at a daily dose of 300 mg affects the frequency of long-term postoperative cardiovascular complications and re-intervention in patients after revascularization operations on the coronary arteries. The second goal is assessing the relationship between the grade monocytes inflammatory response and the level of heteroplasmy of the mitochondrial genome of blood leukocytes with the frequency of cardiovascular complications and re-interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age >40 and <75 years
2. Patients with coronary arteries atherosclerosis for whom coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) is indicated
3. Patients passed a complex of instrumental and laboratory examinations before revascularization, including ECG, echocardiography, visualization of coronary vessels by X-ray contrast angiography, or CT, screening for atherosclerotic lesions of large arteries, including common carotid arteries, abdominal segment of the aorta, arteries of the lower extremities, biochemical analysis of blood included assessment of cholesterol, triglycerides, low density lipoproteins, high density lipoproteins and glucose levels.
4. The possibility of monitoring the patient for 12 months after revascularization, including phone contacts and visits to the clinic after 6 and 12 months.
5. Patient or legal authorized representative capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Repeated revascularization surgery.
2. Critical and urgent cardiovascular conditions: tissue ischemia stage III-IV, stroke, acute coronary syndrome, myocardial infarction, chronic heart failure III and IV class NYHA (New York Heart Association).
3. Other critical and urgent conditions not associated with cardiovascular diseases, including the need for urgent interventions, chronic renal failure stages IV-V (creatinine clearance < 30 ml / min according to the Cockcroft-Gault Equation)
4. High degree of disability of the patient (4 or higher points on the modified Rankin scale).
5. History of systemic autoimmune diseases.
6. Significant weight loss (> 10% of body weight in the previous year) of unknown etiology.
7. Conditions that limit adherence to participation in the study (dementia, neuropsychiatric diseases, drug addiction, alcoholism, etc.).
8. Participation in other clinical studies (or use of investigational substances) within 3 months prior to study entry.
9. Patients with malignant tumors, including the postoperative period with chemotherapy and / or radiation therapy.
10. Carriers of HIV or viral hepatitis
11. Pregnancy or breast feeding
12. Refusal to participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of fatal cardiovascular events | Evaluated in 12 months from revascularisation interventions
  Fatal cardiovascular events include: death from myocardial infarction, other forms of coronary heart disease (CHD), stroke, including sudden death and death within 24 hours of symptom onset, death from other non-coronary cardiovascular diseases except definitely non-atherosclerotic causes of death.
Frequency of clinically significant cardiovascular events | Evaluated in 12 months from revascularisation interventions
  Clinically significant cardiovascular events include: acute myocardial infarction and acute coronary syndrome, acute cerebrovascular accident, progressive heart failure
Frequency of indications for a second revascularization | Evaluated in 12 months from revascularisation interventions

SECONDARY OUTCOMES:
Change in the degree of stenosis of the coronary arteries | Evaluated in 6 and in 12 months from revascularisation interventions
  According to angiography examination
B-mode ultrasound of carotid arteries | Evaluated in 6 and in 12 months from revascularisation interventions
  Variation of intima-media thickness of common carotid arteries
Change in the level of cytokine response of monocytes after double stimulation with lipopolysaccharide in in vitro cell culture | Evaluated in 6 and in 12 months from revascularisation interventions
  Cytokine level measurement by ELISA (TNF-a; IL-1b; IL-6; IL-8; IL-10; CCL2) after the first and second LPS stimulation of monocytes.
Changes in the percentage of heteroplasmy of the mitochondrial genome of blood leukocytes in variants associated with atherosclerosis | Evaluated in 6 and in 12 months from revascularisation interventions
  Includes variants m.12315G>A, m.13513G>A, m.14459G>A, m.14846G>A, m.15059G>A, m.1555A>G, m.3256C>T, m.3336T>C, m.5178C>A, m.652delG measured with quantitative PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Atherosclerosis Research, Moscow, Russia

REFERENCES:
- [Background] Falk E. Pathogenesis of atherosclerosis. J Am Coll Cardiol. 2006 Apr 18;47(8 Suppl):C7-12. doi: 10.1016/j.jacc.2005.09.068. PMID 16631513
- [Background] Bradley JM, Organ CL, Lefer DJ. Garlic-Derived Organic Polysulfides and Myocardial Protection. J Nutr. 2016 Feb;146(2):403S-409S. doi: 10.3945/jn.114.208066. Epub 2016 Jan 13. PMID 26764335
- [Background] Orekhov AN, Tertov VV. In vitro effect of garlic powder extract on lipid content in normal and atherosclerotic human aortic cells. Lipids. 1997 Oct;32(10):1055-60. doi: 10.1007/s11745-997-0136-7. PMID 9358431
- [Background] Orekhov AN, Grunwald J. Effects of garlic on atherosclerosis. Nutrition. 1997 Jul-Aug;13(7-8):656-63. doi: 10.1016/s0899-9007(97)83010-9. PMID 9263259
- [Background] Imaizumi VM, Laurindo LF, Manzan B, Guiguer EL, Oshiiwa M, Otoboni AMMB, Araujo AC, Tofano RJ, Barbalho SM. Garlic: A systematic review of the effects on cardiovascular diseases. Crit Rev Food Sci Nutr. 2023;63(24):6797-6819. doi: 10.1080/10408398.2022.2043821. Epub 2022 Feb 23. PMID 35193446
- [Background] Mollahosseini M, Hosseini-Marnani E, Panjeshahin A, Panbehkar-Jouybari M, Gheflati A, Mozaffari-Khosravi H. A systematic review of randomized controlled trials related to the effects of garlic supplementation on platelet aggregation. Phytother Res. 2022 Nov;36(11):4041-4050. doi: 10.1002/ptr.7556. Epub 2022 Oct 12. PMID 36222178
- [Background] Panyod S, Wu WK, Chen PC, Chong KV, Yang YT, Chuang HL, Chen CC, Chen RA, Liu PY, Chung CH, Huang HS, Lin AY, Shen TD, Yang KC, Huang TF, Hsu CC, Ho CT, Kao HL, Orekhov AN, Wu MS, Sheen LY. Atherosclerosis amelioration by allicin in raw garlic through gut microbiota and trimethylamine-N-oxide modulation. NPJ Biofilms Microbiomes. 2022 Jan 27;8(1):4. doi: 10.1038/s41522-022-00266-3. PMID 35087050
- [Background] Reinhart KM, Talati R, White CM, Coleman CI. The impact of garlic on lipid parameters: a systematic review and meta-analysis. Nutr Res Rev. 2009 Jun;22(1):39-48. doi: 10.1017/S0954422409350003. PMID 19555517
- [Background] Orekhov AN, Sobenin IA, Korneev NV, Kirichenko TV, Myasoedova VA, Melnichenko AA, Balcells M, Edelman ER, Bobryshev YV. Anti-atherosclerotic therapy based on botanicals. Recent Pat Cardiovasc Drug Discov. 2013 Apr;8(1):56-66. doi: 10.2174/18722083113079990008. PMID 23176379
- [Background] Sobenin IA, Pryanishnikov VV, Kunnova LM, Rabinovich YA, Martirosyan DM, Orekhov AN. The effects of time-released garlic powder tablets on multifunctional cardiovascular risk in patients with coronary artery disease. Lipids Health Dis. 2010 Oct 19;9:119. doi: 10.1186/1476-511X-9-119. PMID 20958974
- [Background] Wlosinska M, Nilsson AC, Hlebowicz J, Hauggaard A, Kjellin M, Fakhro M, Lindstedt S. The effect of aged garlic extract on the atherosclerotic process - a randomized double-blind placebo-controlled trial. BMC Complement Med Ther. 2020 Apr 29;20(1):132. doi: 10.1186/s12906-020-02932-5. PMID 32349742
- [Background] Lindstedt S, Wlosinska M, Nilsson AC, Hlebowicz J, Fakhro M, Sheikh R. Successful improved peripheral tissue perfusion was seen in patients with atherosclerosis after 12 months of treatment with aged garlic extract. Int Wound J. 2021 Oct;18(5):681-691. doi: 10.1111/iwj.13570. Epub 2021 Feb 16. PMID 33590955
- [Background] Hamal S, Cherukuri L, Birudaraju D, Matsumoto S, Kinninger A, Chaganti BT, Flores F, Shaikh K, Roy SK, Budoff MJ. Short-term impact of aged garlic extract on endothelial function in diabetes: A randomized, double-blind, placebo-controlled trial. Exp Ther Med. 2020 Feb;19(2):1485-1489. doi: 10.3892/etm.2019.8377. Epub 2019 Dec 27. PMID 32010327
- [Background] Gao X, Xue Z, Ma Q, Guo Q, Xing L, Santhanam RK, Zhang M, Chen H. Antioxidant and antihypertensive effects of garlic protein and its hydrolysates and the related mechanism. J Food Biochem. 2020 Feb;44(2):e13126. doi: 10.1111/jfbc.13126. Epub 2019 Dec 26. PMID 31877235
- [Background] Ried K. Garlic lowers blood pressure in hypertensive subjects, improves arterial stiffness and gut microbiota: A review and meta-analysis. Exp Ther Med. 2020 Feb;19(2):1472-1478. doi: 10.3892/etm.2019.8374. Epub 2019 Dec 27. PMID 32010325
- [Background] Piragine E, Citi V, Lawson K, Calderone V, Martelli A. Potential Effects of Natural H2S-Donors in Hypertension Management. Biomolecules. 2022 Apr 14;12(4):581. doi: 10.3390/biom12040581. PMID 35454169